CLINICAL TRIAL: NCT00537719
Title: A Single-Blind, Randomized, Placebo-Controlled Study in Healthy Men and Women to Determine the Effect of Single Subcutaneous Injections of GSK716155 on Gastric Emptying Time for Solid and Liquid Components of a Meal
Brief Title: Scintigraphy Study to Assess Gastric Emptying in Healthy Subjects Given GSK716155 or Placebo.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLP107030
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: healthy; pharmacodynamics; glucagon-like peptide 1; pharmacokinetics; scintigraphy; radiation; albiglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- GSK716155 (Active Comparator): albiglutide subcutaneous injection
  Interventions: Drug: GSK716155
- placebo (Placebo Comparator): placebo injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK716155 — albiglutide subcutaneous injection
  Arms: GSK716155
Drug: Placebo — placebo injection
  Other Names: GSK716155
  Arms: placebo

SUMMARY:
This study will use scintigraphy techniques to measure gastric emptying rate of liquid and solid food at baseline and after administration of GSK716155 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women, between the ages of 18 and 65, and have a Body Mass Index (BMI) of between 20 and 32.
* If female, the subject must be not be capable of having children.

Exclusion Criteria:

* Subjects must not use tobacco, nicotine, or illegal drugs of abuse, and must not take caffeine or alcohol for 24 hours before dosing and before each set of scintigraphy procedures.
* Subjects may not have HIV, hepatitis, elevated fasting blood sugar levels, high blood pressure, heart, lung, liver, gall bladder, gastrointestinal, pancreatic, or kidney disease, or untreated thyroid disease.
* Subjects must not have a history of alcohol abuse, must not take prescription or non-prescription drugs within 7 days of Day 1 and Day 8 of the study, and must not have previous exposure to any GLP-1 mimetic or exenatide.
* Prior radiation exposures must meet certain limits in order to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-12-07 (Actual); Primary Completion 2008-04-04 (Actual); Study Completion 2008-04-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the time to 50% gastric emptying (gastric emptying t½) of the solid and liquid components of a meal at 72 hours after dosing in healthy volunteers. | 3 Days

SECONDARY OUTCOMES:
Exploratory correlation of % contents remaining in stomach after a meal.GSK716155 concentration before meal & at the time gastric emptying is complete. Safety and tolerability parameters each visit. | 3 Days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study GLP107030 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/GLP107030?search=study&study_ids=GLP107030#rs
- Available data/document: Individual Participant Data Set: GLP107030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: GLP107030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: GLP107030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: GLP107030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: GLP107030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: GLP107030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: GLP107030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register